CLINICAL TRIAL: NCT03682354
Title: Erector Spinae Plane Block Versus Intercostal Nerve Block Combined With Patient-controlled Intravenous Analgesia in Video-assisted Thoracic Surgery
Brief Title: ESPB Versus INB With PCIA in Video-assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2018123
Record Dates: First submitted 2018-08-26; First posted 2018-09-24 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Lung Diseases
Keywords: Erector spinae plane block; Video-assisted thoracic surgery;; Intercostal nerve block; Patient-controlled intravenous analgesia
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal Nerve Block with PCIA (Active Comparator): Intercostal Nerve Block with patient-controlled intravenous analgesia
  Interventions: Drug: Intercostal Nerve Block with PCIA
- Erector Spinae Plane Block (ESPB) (Experimental): Continuous Erector Spinae Plane Block
  Interventions: Drug: Erector Spinae Plane Block (ESPB)

INTERVENTIONS:
Drug: Intercostal Nerve Block with PCIA — Intercostal nerve block consists in the injection of Ropivacaine (4 ml,0.5%) in related intercostal spaces. Patient-controlled intravenous analgesia regimen is conducted with sufentanil.
  Arms: Intercostal Nerve Block with PCIA
Drug: Erector Spinae Plane Block (ESPB) — Erector Spinae Plane Block consists in the injection of Ropivacaine (20ml, 0.5%), in the anatomical plane between the Erector Spinae muscles and transverse process, laterally to the spinous process of T5 . The catheter was inserted and secured in place under ecographic guidance, and a patient-controlled regional anesthesia regimen was conducted with 0.2% ropivacaine.
  Arms: Erector Spinae Plane Block (ESPB)

SUMMARY:
A randomized prospective trial to test the non-inferiority of erector spinae plane block (ESPB) in comparison with intercostal nerve block combined with patient-controlled intravenous analgesia in Thoracoscopic lung surgery

DETAILED DESCRIPTION:
For patients undergoing thoracic surgery, postoperative pain greatly limited their recovery.Multimodal analgesia have shown good efficacy but without reaching full pain relief.

The primary goal of this study is to observe the effect of ultrasound-guided erector spinae plane block in comparison with intercostal nerve block combined with patient-controlled intravenous analgesia in video assisted thoracic lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients to receive video assisted thoracoscopic lobectomy or bullectomy .

Exclusion Criteria:

* 1. Patient refusal 2. Heavy skin eruption and infection at site of injection. 3. Coagulopathy. 4. Allergy to local anesthetics. 5. Taking analgesics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Pain score (NRS) | 4 hours from the end of procedure
  Numeric Rating Scale is an 11-point scale used by doctors to evaluate patients' pain, where 0 is no pain and 10 the worst imaginable pain. For postoperative patients, an higher score shows inadequate analgesia and worse outcome.

SECONDARY OUTCOMES:
Pain score (NRS) | 8, 24,48 hours from the end of procedure
  Numeric Rating Scale is an 11-point scale used by doctors to evaluate patients' pain, where 0 is no pain and 10 the worst imaginable pain. For postoperative patients, an higher score shows inadequate analgesia and worse outcome.
Analgesics consumption | During operation,4, 8, 24,48 hours from the end of procedure
  Analgesics include opioids and nonsteroidal anti-inflammatory drugs
Incidence of side effects and complication during study | During operation,4, 8, 24,48 hours from the end of procedure
  Side effects and complication

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang T, Wang X, Yu Z, Li M. Programmed Intermittent Bolus for Erector Spinae Plane Block Versus Intercostal Nerve Block With Patient-controlled Intravenous Analgesia in Video-assisted Thoracoscopic Surgery: A Randomized Controlled Noninferiority Trial. Clin J Pain. 2024 Feb 1;40(2):99-104. doi: 10.1097/AJP.0000000000001174. PMID 37975501